CLINICAL TRIAL: NCT01248819
Title: Double Blind Randomized Phase III Controlled Trial Comparing the Effect of Intraperitoneal Nebulization of Ropivacaine With Intraperitoneal Instillation of Ropivacaine on Pain Control After Laparoscopic Cholecystectomy
Brief Title: Local Anesthetic Nebulization and Instillation for Pain Control After Laparoscopic Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: San Gerardo Hospital (Other)
Collaborators: Hôpital de Hautepierre (Other)
Responsible Party: Pablo M Ingelmo, MD, First Service of anesthesia and intensive care. San Gerardo Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AR HSG 04-2008
Record Dates: First submitted 2010-11-24; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2008-03

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Laparoscopic Cholecystectomy; Nebulization; Ropivacaine
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Instillation (Active Comparator): Instillation of Ropivacaine 100 mg in the abdominal cavity
  Interventions: Drug: Ropivacaine 100 mg
- Nebulization (Experimental): Nebulization of Ropivacaine 60 mg in the abdominal cavity
  Interventions: Drug: Ropivacaine 60 mg

INTERVENTIONS:
Drug: Ropivacaine 60 mg — Nebulization grou received intraperitoneal instillation of saline 20 ml on the gall bladder after induction of pneumoperitoneum but before dissection of gall bladder plus intraperitoneal nebulization of ropivacaine 1% 3 ml (30 mg) the start of gall bladder dissection and again at the end of surgery just before deflation of pneumoperitoneum (total of 60 mg). The first ropivacaine nebulization was performed over 5-6 minutes using the Aeroneb Pro® device through the umbilical port while the other ports were being inserted, while second nebulization was performed before the withdrawal of the ports
  Arms: Nebulization
Drug: Ropivacaine 100 mg — Instillation group received intraperitoneal instillation of ropivacaine 0.5%, 20 ml (100 mg) on the gall bladder after induction of pneumoperitoneum but before dissection of gall bladder plus and intraperitoneal nebulization of normal saline 3 ml before the start of gall bladder dissection and again at the end of surgery just before deflation of pneumoperitoneum. The first saline nebulization was performed over 5-6 minutes using the Aeroneb Pro® device through the umbilical port while the other ports were being inserted, while second nebulization was performed before the withdrawal of the ports
  Arms: Instillation

SUMMARY:
Studies evaluating intraperitoneal local anesthetic instillation for pain relief after laparoscopic procedures have provided conflicting results. This randomized, double-blind study was designed to assess the effects of a novel intraperitoneal local anesthetic administration technique using nebulization on pain relief after laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Studies evaluating intraperitoneal local anesthetic (LA) instillation for pain relief after laparoscopic cholecystectomy have provided conflicting results. One of the factors that might contribute to failure of the instillation technique may be related to inadequate distribution of local anesthetic throughout the peritoneal surface. In contrast, nebulization should provide a uniform spread of drugs throughout the peritoneal cavity and thus may be beneficial to improve pain relief after laparoscopic procedures. A recent study reported that bupivacaine nebulization significantly reduced pain after laparoscopic cholecystectomy compared with bupivacaine instillation in the gallbladder bed. However, these investigators used a custom-made nebulization system that needs a separate gas source and tubing that is cumbersome and may not be easily available.

Recently, the investigators reported that a microvibration-based nebulization device (Aeroneb Pro® system, Aerogen, Galway, Ireland) could be used for ropivacaine delivery into the insufflation gas required to create pneumorpeitoneum. The investigators hypothesized that intraperitoneal ropivacaine nebulization would provide superior pain relief after laparoscopic cholecystectomy than intraperitoneal ropivacaine instillation. This randomized, double blind, controlled clinical trial was designed to assess the analgesic efficacy of ropivacaine nebulization using the Aeroneb Pro® device laparoscopic cholecystectomy compared with intraperitoneal ropivacaine instillation.

ELIGIBILITY:
Inclusion Criteria:

* ASA Score I-III
* Scheduled for laparoscopic cholecystectomy
* Free from pain in preoperative period
* Not using analgesic drugs before surgery
* Without cognitive impairment or mental retardation
* Written informed consent

Exclusion Criteria:

* Emergency/urgency surgery
* Postoperative admission in an intensive care unit
* Cognitive impairment or mental retardation
* Progressive degenerative diseases of the CNS
* Seizures or chronic therapy with antiepileptic drugs
* Severe hepatic or renal impairment
* Pregnancy or lactation
* Allergy to one of the specific drugs under study
* Acute infection or inflammatory chronic disease
* Alcohol or drug addiction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-04; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain | 48 hours
  Postoperative pain was assessed by Visual analgue scale (VAS 0 to 100 points) at rest (static VAS) and after a deep inspiration or cough (dynamic VAS). The proportion of patients with adequate pain control after surgery (dynamic VAS < 3) will also be assessed.

SECONDARY OUTCOMES:
Morphine consumption (mg) | Up to 48 hours
  The total dose of morphine at every evaluation after awakening will be quantified using the PACU clinical chart and/or PCA infusers memory display
Time of unassisted walking | Up to 48 hours
  Unassisted walking time is defined as the time in hours between PACU discharge and when the patient is able to walk out of his room and back to bed without any assistance.
Hospital morbidity | Up to 48 hours
  All complications or adverse effects associated or possibly associated with the interventions under study, surgery or anesthesia will be quantified using the anesthesia charts, surgical charts, surgical database.
Time to hospital discharge | 48 hours
  We define hospital stay as the elapsed time between surgery and hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Pablo M Ingelmo, MD, Principal Investigator — San Gerardo Hospital
Locations (1):
- San Gerardo Hospital, Monza, MB, Italy

REFERENCES:
- [Result] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268
- [Result] Greib N, Schlotterbeck H, Dow WA, Joshi GP, Geny B, Diemunsch PA. An evaluation of gas humidifying devices as a means of intraperitoneal local anesthetic administration for laparoscopic surgery. Anesth Analg. 2008 Aug;107(2):549-51. doi: 10.1213/ane.0b013e318176fa1c. PMID 18633034
- [Result] Schlotterbeck H, Schaeffer R, Dow WA, Diemunsch P. Cold nebulization used to prevent heat loss during laparoscopic surgery: an experimental study in pigs. Surg Endosc. 2008 Dec;22(12):2616-20. doi: 10.1007/s00464-008-9841-z. Epub 2008 Mar 18. PMID 18347861